CLINICAL TRIAL: NCT03859778
Title: Evaluation of Pharmacy Students' Perception of Opioid / Opiate Dependence: Cross-sectional National Study
Brief Title: Evaluation of Pharmacy Students' Perception of Opioid / Opiate Dependence
Acronym: STUD_TOX
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UFR Pharmacie (Clermont-Ferrand) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-427
Record Dates: First submitted 2019-02-21; First posted 2019-03-01 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-02

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid-Related Disorders; student; Community Pharmacy Services
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pharmacy students
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — French pharmacy students will be contacted by email thanks to the student associations and scolarity departments. Answer to the survey will be done online

SUMMARY:
The pharmacist in his professional activity may have to manage opioid dependent patients. This professional activity will result in the provision of opioid substitution treatment (OST), single-use syringes, harm reduction kits and a prevention advice for the reduction of toxicity and infection risks.

Since the 1990s, the consumption of OST has been steadily increasing. According to the OFDT (French Observatory of Drugs and Drug Addiction), the number of patients under OST is about 150 000 patients. Since high-dose buprenorphine is prescribed for approximately two-thirds of patients, it remains the most frequently prescribed OST in France.

Recently, a French association assisting drug users (ASUD - Auto-support des usagers de drogues) performed a study in Paris (20/07/2018 - 25/08/2018) to assess the delivery of opioid replacement therapies by community pharmacists. In this study, 71% of pharmacists refused to deliver opioid replacement therapies. The main reasons reported were security (56%) and activity saturation, meaning that pharmacists considered that they had too many patients using opioid drugs. In France, the refusal of a pharmacist to deliver drugs is a punishable offence. According to the Code of ethics of pharmacists, pharmacists must respect life and people without discrimination. Pharmacists have a low perception of patients suffering from opioid addiction. Another study performed by ASUD in 93 community pharmacies, showed that pharmacists used the term "toxicomaniacs" instead of "drug users". Most pharmacists had had a bad experience with drugs users, with physical and verbal aggressions. The conclusions of this study showed that pharmacists lacked knowledge of drug users and drug use. Pharmacists knew about harm reduction kits for opioid users (containing sterile syringes, needles, water, antiseptics, etc.) and had already opened them, but very few knew how to use them. More worryingly, some pharmacists did not understand the harm reduction strategies available It thus appears that community pharmacists have a difficult relationship with opioid-dependent patients, even though these pharmacists have received education in the management of addictions during their studies. Indeed, it can consider that these courses should help to better understand the addictive disease both in its nosological / semiological and therapeutic components. Thus, it would be interesting to evaluate the impact of addiction education on pharmacists' perception of opioid dependence. In this perspective, it would be interesting to focus on pharmacy students.

The objective of this study will be to evaluate the perception by pharmacy students of opioid dependent patients. Investigator would like to know if pharmacy students consider opioid addiction to be an illness and whether having taken education on drug use and addictions changes this perception.

DETAILED DESCRIPTION:
This observational and cross-sectional study will be conducted as a survey using the REDCap software and the response to this survey will be done online, in real time, with an automatic, secure and centralized data collection (CHU Clermont-Ferrand).

French pharmacy students will be contacted by email thanks to the student associations and scolarity departments. Answer to the survey will be done online.

ELIGIBILITY:
Inclusion Criteria:

* French pharmacy students

Exclusion Criteria:

* Age <18 years
* Other health students
* Graduated pharmacist
* First year pharmacy student

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French pharmacy students
Sampling Method: Non-Probability Sample
Enrollment: 2034 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Perception of opioid / opiate dependence as a disease | At day 1
  visual analogic scale: -10 (it is not a disease), 0 (neutral) and +10(it is a disease)

SECONDARY OUTCOMES:
Proportion of courses on drug addiction during pharmacy studies | At day 1
  yes/no (percentage)
Study year of courses on drug addiction during pharmacy studies | At day 1
  2nd, 3rd, 4th, 5th and/or 6th year of study in pharmacy
Perception of the pharmacist's missions on the dispensing of opioid substitution treatments (buprenorphine and methadone) and harm reduction kit / single use syringe | At day 1
  visual analogic scale: -10 (it's not normal), 0 (neutral) and +10 (it's normal)
Perception of the efficacy of opioid substitution treatments (buprenorphine and methadone) | At day 1
  visual analogic scale: -10 (it is not effective), 0 (neutral) and +10 (it is effective)
Proportion of realization of internships or temporary employment in pharmacy | At day 1
  yes / no (percentage)
Proportion of delivery of opioid substitution treatments (buprenorphine and methadone) | At day 1
  yes / no (percentage)
Proportion of tobacco (cigarettes) use | At day 1
  yes / no (percentage)
Proportion of electronic cigarettes use | At day 1
  yes / no (percentage)
Proportion of alcohol use | At day 1
  yes / no (percentage)
Proportion of alcohol use (>10 alcohol units per week) | At day 1
  yes / no (percentage)
Proportion of cannabis use | At day 1
  yes / no (percentage)
Frequency of cannabis use (for users) | At day 1
  Daily, weekly, monthly, occasional or experimentation
Proportion of personal experience with a relative having or having had a problem of drug use | At day 1
  yes / no (percentage)
Academic year in pharmacy at the time of the answer | At day 1
  2nd / 3rd / 4th / 5th / 6th year of study in pharmacy
Estimation of attendance to courses | At day 1
  Visual analogic scale: 0 (no attendance) - 100 (full attendance)
Estimation of annual average mark during the past university year | At day 1
  <10, 10-12, 12-14, 14-16 and >16/20
Demographic information | At day 1
  age and sex

CONTACTS AND LOCATIONS:
Overall Officials: David BALAYSSAC, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France